CLINICAL TRIAL: NCT00985725
Title: Phase 2, Multicenter, Randomized, Double-blind, Placebo-Controlled, Study to Evaluate the Efficacy, Safety, and Tolerability of SPD489 in Adults With Clinically Significant, Persistent Executive Function Impairments (EFI) and Partial or Full Remission of Recurrent Major Depressive Disorder
Brief Title: SPD489 in Adults With Persistent Executive Function Impairments (EFI) and Partial or Full Remission of Recurrent Major Depressive Disorder
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Shire (Industry)
Responsible Party: Sponsor
Organization: Takeda (Industry)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: SPD489-205
Record Dates: First submitted 2009-09-25; First posted 2009-09-28 (Estimated); Results first posted 2012-04-06 (Estimated); Last update posted 2021-06-08 (Actual); Status verified 2021-05

CONDITIONS: Major Depressive Disorder
Keywords: Major Depressive Disorder
MeSH Terms: conditions — Depressive Disorder, Major | interventions — Lisdexamfetamine Dimesylate

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Active (Experimental): SPD489
  Interventions: Drug: SPD489 (Lisdexamfetamine dimesylate)
- Placebo (Placebo Comparator): Placebo
  Interventions: Drug: Matching placebo

INTERVENTIONS:
Drug: SPD489 (Lisdexamfetamine dimesylate) — Oral, 20, 30, 40, 50, 60, and 70mg capsules, once daily
  Other Names: Vyvanse
  Arms: Active
Drug: Matching placebo — oral, once daily
  Arms: Placebo

SUMMARY:
To evaluate the efficacy of SPD489 for the treatment of executive function impairments (EFI) when used as an adjunct to stable, standard therapy in the setting of partial or full remission from recurrent Major Depressive Disorder (MDD) as measured by the Global Executive Composite (GEC) T-score of the Behavioral Rating Inventory of Executive Functioning - Adult Version (BRIEF-A).

ELIGIBILITY:
Inclusion Criteria:

* Adults aged 18-55 with a primary diagnosis of nonpsychotic uni-polar depression

Exclusion Criteria:

* Current co-morbid psychiatric disorder

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 143 (Actual)
Dates: Start 2009-10-29 (Actual); Primary Completion 2011-04-18 (Actual); Study Completion 2011-04-18 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Study Director, Study Director — Takeda
Locations (33):
- United States (33):
  - Sun Valley Research Center, Imperial, California
  - Pharmacology Research Center, Los Alamitos, California
  - Excell Research, Oceanside, California
  - Neuropsychiatric Resesarch Center of Orange County, Santa Ana, California
  - Connecticut Clincal Research, Cromwell, Connecticut
  - Clinical Neuroscience Solutions, Inc., Jacksonville, Florida
  - Amit Vijapura, MD, Jacksonville, Florida
  - Scientific Clinical Research, Inc., North Miami, Florida
  - Clinical Neuroscience Solutions, Inc., Orlando, Florida
  - Atlanta Institute of Medicine & Research, Atlanta, Georgia
  - Carman Research, Smyrna, Georgia
  - Joliet Center for Clinical Research, Joliet, Illinois
  - Capstone Clinical Research, Libertyville, Illinois
  - Psychiatric Associates, Overland Park, Kansas
  - AccelRx Research, Fall River, Massachusetts
  - St. Charles Psychiatric Associates, Saint Charles, Missouri
  - PsychCare Consultants Research, St Louis, Missouri
  - Premier Psychiatric Research Institute, LLC, Lincoln, Nebraska
  - Richmond Behavioral Associates, Staten Island, New York
  - North Carolina Neuropsychiatry, PA, Chapel Hill, North Carolina
  - Duke University Medical Center, Durham, North Carolina
  - Richard H. Weisler, MD, PA & Associates, Raleigh, North Carolina
  - Patient Priority Clinical Sites, LLC, Cincinnati, Ohio
  - Lehigh Center for Clinical Research, Allentown, Pennsylvania
  - Paramount Clinical Research, Bridgeville, Pennsylvania
  - Suburban Research Associates, Media, Pennsylvania
  - FutureSearch Trials of Dallas, LP, Dallas, Texas
  - Bayou City Resesarch, LTD, Houston, Texas
  - Red Oak Psychiatry Associates, PA, Houston, Texas
  - University Hills Clinical Research, Irving, Texas
  - R/D Clinical Research, Inc., Lake Jackson, Texas
  - Wharton Research Center, Wharton, Texas
  - Northwest Clinical Research Center, Bellevue, Washington

REFERENCES:
- [Derived] Madhoo M, Keefe RS, Roth RM, Sambunaris A, Wu J, Trivedi MH, Anderson CS, Lasser R. Lisdexamfetamine dimesylate augmentation in adults with persistent executive dysfunction after partial or full remission of major depressive disorder. Neuropsychopharmacology. 2014 May;39(6):1388-98. doi: 10.1038/npp.2013.334. Epub 2013 Dec 6. PMID 24309905

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Subjects clinically stable on an anti-depressant were randomized (1:1) to LDX or placebo augmentation for 9 weeks. Double-blind LDX or placebo was administered orally as adjunctive therapy (20 to 70 mg per day, titrated over the initial 6 weeks), with the optimal individual dose being continued during a 3-week dose maintenance period.
Groups:
- Lisdexamfetamine Dimesylate (LDX): Lisdexamfetamine Dimesylate (LDX, SPD489) is administered orally once-daily at doses of either 20, 30, 40, 50, 60, or 70 mg for 9 weeks.
- Placebo: Administered orally once-daily for 9 weeks.
Period: Overall Study
Arm/Group | Lisdexamfetamine Dimesylate (LDX) | Placebo
Started | 71 | 72
Completed | 60 | 59
Not Completed | 11 | 13
Not completed — Adverse Event | 4 | 1
Not completed — Protocol Violation | 1 | 3
Not completed — Withdrawal by Subject | 4 | 4
Not completed — Lost to Follow-up | 1 | 1
Not completed — Lack of Efficacy | 0 | 1
Not completed — Non-compliance | 1 | 2
Not completed — Out-of-window visits | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Lisdexamfetamine Dimesylate (LDX) | Placebo | Total
Number analyzed (Participants) | 71 | 72 | 143
Age, Continuous [Mean (Standard Deviation); unit: years] | 41.9 (9.79) | 39.5 (10.59) | 40.7 (10.23)
Age, Customized [Count of Participants; unit: Participants]
  18 to 39 years | 28 | 34 | 62
  40 to 55 years | 43 | 38 | 81
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 51 | 48 | 99
  Male | 20 | 24 | 44
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 71 | 72 | 143

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Behavior Rating Inventory of Executive Function - Adult Version Global Executive Composite T-score (BRIEF-A GEC T) at Week 9, Last Observation Carried Forward (LOCF)
Description: BRIEF-A Global Executive Composite assesses behavioral aspects of executive function. Items are rated 1 (never), 2 (sometimes), and 3 (often). There is no range for a total score. Raw scale scores are used to generate T-scores. A reduction in score indicates less impairment.
Time Frame: Baseline and week 9
Population: The Full Analysis Set (FAS) defined as all randomized subjects who took at least 1 dose of randomized investigational product and had at least 1 primary efficacy assessment after baseline.
Measure: Least Squares Mean (Standard Error); unit: T-scores
Arm/Group | Lisdexamfetamine Dimesylate (LDX) | Placebo
Number analyzed (Participants) | 71 | 72
T-scores | -21.2 (1.67) | -13.2 (1.66)
Statistical Analysis 1: Comparison: Lisdexamfetamine Dimesylate (LDX) vs Placebo; Test type: Superiority or Other; p = 0.0009, ANCOVA; Mean Difference (Final Values) = -8.0, 95% CI 2-sided [-12.7 to -3.3]

2. Secondary Outcome: Change From Baseline in Montgomery-Ǻsberg Depression Rating Scale (MADRS) Total Score at Week 9 - (LOCF)
Description: MADRS is a validated, 10-item rating scale with each item being scored on a scale from 0-6 with a total score ranging from 0-60. Lower scores indicate a decreased severity of depression.
Time Frame: Baseline and week 9
Population: FAS
Measure: Least Squares Mean (Standard Error); unit: Scores on a scale
Arm/Group | Lisdexamfetamine Dimesylate (LDX) | Placebo
Number analyzed (Participants) | 71 | 72
Scores on a scale | -5.0 (0.66) | -3.1 (0.66)
Statistical Analysis 1: Comparison: Lisdexamfetamine Dimesylate (LDX) vs Placebo; Test type: Superiority or Other; p = 0.0465, ANCOVA; Mean Difference (Final Values) = -1.9, 95% CI 2-sided [-3.7 to 0.0]

3. Secondary Outcome: Change From Baseline in BRIEF-A T-scores at Week 9, LOCF
Description: BRIEF-A is a validated 75-item questionnaire. Items are rated 1 (never), 2 (sometimes), and 3 (often). There is no range for a total score. Raw scale scores are used to generate T-scores. A reduction in score indicates less impairment.
Time Frame: Baseline and week 9
Population: FAS
Measure: Least Squares Mean (Standard Error); unit: T-scores
Arm/Group | Lisdexamfetamine Dimesylate (LDX) | Placebo
Number analyzed (Participants) | 71 | 72
T-scores
  Behavioral recognition index | -17.4 (1.51) | -12.3 (1.50)
  Inhibit subscale | -13.5 (1.26) | -9.3 (1.25)
  Shift subscale | -16.2 (1.51) | -10.6 (1.50)
  Emotional control subscale | -13.8 (1.48) | -10.1 (1.47)
  Self-monitor subscale | -13.8 (1.36) | -10.7 (1.35)
  Metacognition index | -21.1 (1.67) | -12.2 (1.66)
  Initiate subscale | -19.4 (1.57) | -10.8 (1.56)
  Working memory subscale | -20.1 (1.65) | -11.0 (1.64)
  Plan/Organize subscale | -18.7 (1.58) | -11.3 (1.57)
  Task monitor subscale | -16.8 (1.63) | -11.9 (1.62)
  Organization of materials subscale | -15.2 (1.49) | -8.2 (1.48)
Statistical Analysis 1: Comparison: Lisdexamfetamine Dimesylate (LDX) vs Placebo; Behavioral recognition index; Test type: Superiority or Other; p = 0.0181, ANCOVA; Mean Difference (Final Values) = -5.1, 95% CI 2-sided [-9.4 to -0.9]
Statistical Analysis 2: Comparison: Lisdexamfetamine Dimesylate (LDX) vs Placebo; Inhibit subscale; Test type: Superiority or Other; p = 0.0204, ANCOVA; Mean Difference (Final Values) = -4.2, 95% CI 2-sided [-7.7 to -0.7]
Statistical Analysis 3: Comparison: Lisdexamfetamine Dimesylate (LDX) vs Placebo; Shift subscale; Test type: Superiority or Other; p = 0.0090, ANCOVA; Mean Difference (Final Values) = -5.6, 95% CI 2-sided [-9.8 to -1.4]
Statistical Analysis 4: Comparison: Lisdexamfetamine Dimesylate (LDX) vs Placebo; Emotional control subscale; Test type: Superiority or Other; p = 0.0793, ANCOVA; Mean Difference (Final Values) = -3.7, 95% CI 2-sided [-7.9 to 0.4]
Statistical Analysis 5: Comparison: Lisdexamfetamine Dimesylate (LDX) vs Placebo; Self-monitor subscale; Test type: Superiority or Other; p = 0.1014, ANCOVA; Mean Difference (Final Values) = -3.2, 95% CI 2-sided [-7.0 to 0.6]
Statistical Analysis 6: Comparison: Lisdexamfetamine Dimesylate (LDX) vs Placebo; Metacognition index; Test type: Superiority or Other; p = 0.0002, ANCOVA; Mean Difference (Final Values) = -9.0, 95% CI 2-sided [-13.7 to -4.3]
Statistical Analysis 7: Comparison: Lisdexamfetamine Dimesylate (LDX) vs Placebo; Initiate subscale; Test type: Superiority or Other; p = 0.0002, ANCOVA; Mean Difference (Final Values) = -8.6, 95% CI 2-sided [-12.9 to -4.2]
Statistical Analysis 8: Comparison: Lisdexamfetamine Dimesylate (LDX) vs Placebo; Working memory subscale; Test type: Superiority or Other; p = 0.0001, ANCOVA; Mean Difference (Final Values) = -9.1, 95% CI 2-sided [-13.7 to -4.5]
Statistical Analysis 9: Comparison: Lisdexamfetamine Dimesylate (LDX) vs Placebo; Plan/Organize subscale; Test type: Superiority or Other; p = 0.0010, ANCOVA; Mean Difference (Final Values) = -7.5, 95% CI 2-sided [-11.9 to -3.1]
Statistical Analysis 10: Comparison: Lisdexamfetamine Dimesylate (LDX) vs Placebo; Task monitor subscale; Test type: Superiority or Other; p = 0.0357, ANCOVA; Mean Difference (Final Values) = -4.9, 95% CI 2-sided [-9.4 to -0.3]
Statistical Analysis 11: Comparison: Lisdexamfetamine Dimesylate (LDX) vs Placebo; Organization of materials subscale; Test type: Superiority or Other; p = 0.0012, ANCOVA; Mean Difference (Final Values) = -7.0, 95% CI 2-sided [-11.1 to -2.8]

4. Secondary Outcome: Change From Baseline in Central Nervous System Vital Signs Computerized Cognitive Testing Battery Neurocognitive Domain and Index Scores at up to 9 Weeks/Endpoint
Description: This measures the speed and accuracy of basic mental functions. Scores are normalized from raw scores and present an age matched score relative to other people in a normative sample. Scores are normalized with a mean of 100 and standard deviation of 15. Scores < 70 indicate likely deficit and impairment, and scores > 110 indicate high function and capacity. Higher scores are better.
Time Frame: Baseline and up to 9 weeks/Endpoint
Population: FAS
Measure: Mean (Standard Deviation); unit: Response scores
Arm/Group | Lisdexamfetamine Dimesylate (LDX) | Placebo
Number analyzed (Participants) | 71 | 72
Response scores
  Complex information speed processing index | 8.7 (10.13) | 3.7 (9.02)
  Executive function index | 11.0 (14.80) | 6.0 (14.43)
  Neurocognitive index | 11.5 (17.14) | 2.5 (13.74)

5. Secondary Outcome: Percent of Participants With Clinical Global Impression - Severity of Illness (CGI-S) at Baseline
Description: CGI-S assesses the severity of the subject's condition on a 7-point scale ranging from 1 (normal, not at all ill) to 7 (among the most extremely ill)
Time Frame: Baseline
Population: FAS
Measure: Number; unit: percentage of participants
Arm/Group | Lisdexamfetamine Dimesylate (LDX) | Placebo
Number analyzed (Participants) | 71 | 72
percentage of participants
  Normal, not at all ill | 0.0 | 2.8
  Borderline mentally ill | 7.0 | 8.3
  Mildly ill | 42.3 | 36.1
  Moderately ill | 45.1 | 48.6
  Markedly ill | 4.2 | 4.2
  Severely ill | 1.4 | 0.0
  Among the most extremely ill | 0.0 | 0.0

6. Secondary Outcome: Percent of Participants With CGI-S at up to 9 Weeks/Endpoint
Description: as for outcome 5
Time Frame: Up to 9 weeks/Endpoint
Population: FAS population was used for this assessment. However, not all subjects from the FAS completed this assessment, therefore the total number of subjects analyzed for this outcome is less than the total number of subjects that comprise the FAS population.
Measure: Number; unit: percentage of participants
Arm/Group | Lisdexamfetamine Dimesylate (LDX) | Placebo
Number analyzed (Participants) | 69 | 69
percentage of participants
  Normal, not at all ill | 21.7 | 15.9
  Borderline mentally ill | 40.6 | 23.2
  Mildly ill | 20.3 | 24.6
  Moderately ill | 14.5 | 34.8
  Markedly ill | 2.9 | 1.4
  Severely ill | 0.0 | 0.0
  Among the most extremely ill | 0.0 | 0.0

7. Secondary Outcome: Percentage of Participants With Improvement on Clinical Global Impression-Improvement (CGI-I) at Week 9, LOCF
Description: Clinical Global Impression-Improvement (CGI-I) consists of a 7-point scale ranging from 1 (very much improved) to 7 (very much worse). Improvement is defined as a score of 1 (very much improved) or 2 (much improved) on the scale.
Time Frame: Week 9
Population: FAS
Measure: Number; unit: percentage of participants
Arm/Group | Lisdexamfetamine Dimesylate (LDX) | Placebo
Number analyzed (Participants) | 71 | 72
percentage of participants | 60.6 | 38.9

8. Secondary Outcome: Change From Baseline in Endicott Work Productivity Scale (EWPS) Total Score at up to 9 Weeks/Endpoint
Description: The EWPS quantifies work performance, productivity attitudes and behaviors assessing 25 items on a scale ranging from 0 (high performance) to 4 (lowest performance). Scores range from 0 to 100 with 100 representing lowest productivity.
Time Frame: Baseline and up to 9 weeks/Endpoint
Population: as for outcome 6
Measure: Least Squares Mean (Standard Error); unit: Scores on a scale
Arm/Group | Lisdexamfetamine Dimesylate (LDX) | Placebo
Number analyzed (Participants) | 46 | 43
Scores on a scale | -20.4 (2.24) | -15.9 (2.32)
Statistical Analysis 1: Comparison: Lisdexamfetamine Dimesylate (LDX) vs Placebo; Test type: Superiority or Other; p = 0.1731, ANCOVA; Mean Difference (Final Values) = -4.4, 95% CI 2-sided [-10.9 to 2.0]

9. Secondary Outcome: Change From Baseline in Changes in Sexual Functioning Questionnaire (CSFQ-14) Total Scores for Males at Week 9, LOCF
Description: This is a 14 item self-report tool that evaluates sexual functioning. Each item is scored on a 5-point Likert scale ranging from 1 (never) to 5 (always) with total scores ranging from 14 to 70. Higher scores reflect better sexual functioning.
Time Frame: Baseline and week 9
Population: The Safety Analysis Set (SAS) defined as all randomized subjects who took at least 1 dose of investigational product and for whom at least 1 follow-up safety assessment was completed. Only the males from the SAS population were used and not all of them completed this outcome assessment.
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | Lisdexamfetamine Dimesylate (LDX) | Placebo
Number analyzed (Participants) | 20 | 21
Scores on a scale | 2.5 (4.61) | 2.4 (5.34)

10. Secondary Outcome: Change From Baseline in CSFQ-14 Total Scores for Females at Week 9, LOCF
Description: as for outcome 9
Time Frame: Baseline and week 9
Population: Only the females from the SAS population were used and not all of them completed this outcome assessment.
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | Lisdexamfetamine Dimesylate (LDX) | Placebo
Number analyzed (Participants) | 48 | 46
Scores on a scale | 2.7 (8.47) | 1.6 (5.60)

11. Secondary Outcome: Change From Baseline in Short Form-12 Health Survey (SF-12) Scale Total Scores at Week 9
Description: The SF-12 is a 12-item self-report questionnaire that is a subset of the SF-36 Health Survey. The survey captures physical and mental health. Each of the 12 items is scored using various scales with a total score ranging from 0 (lowest level of health) to 100 (highest level of health).
Time Frame: Baseline and week 9
Population: as for outcome 6
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | Lisdexamfetamine Dimesylate (LDX) | Placebo
Number analyzed (Participants) | 66 | 66
Scores on a scale
  Aggregate physical | -0.10 (0.461) | -0.23 (0.473)
  Aggregate mental | 0.69 (0.987) | 0.63 (0.807)

12. Secondary Outcome: Change From Baseline in Quality of Life Enjoyment and Satisfaction Questionnaire (Q-LES-Q) Total Scores at up to 9 Weeks/Endpoint
Description: The Q-LES-Q is a 93-item self-report questionnaire on quality of life and health. Each item is rated on a 5-point scale from 1 (very poor) to 5 (very good) with a total score ranging from 93 to 465. Higher scores indicate greater satisfaction.
Time Frame: Baseline and up to 9 weeks/Endpoint
Population: as for outcome 6
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | Lisdexamfetamine Dimesylate (LDX) | Placebo
Number analyzed (Participants) | 68 | 69
Scores on a scale
  Physical health activities | 17.9 (20.03) | 8.2 (16.82)
  Overall life satisfaction | 12.1 (25.37) | 9.1 (22.27)

13. Secondary Outcome: Change From Baseline in Amphetamine Cessation Symptom Assessment (ACSA) Total Score at Week 11
Description: ACSA scale has 16 symptom items rated on a scale from 0 (not at all) to 4 (extremely) with a possible total score range of 0 to 64. Higher scores indicate greater withdrawal symptom severity.
Time Frame: Baseline and week 11
Population: SAS population was used for this assessment. However, not all subjects from the SAS completed this assessment, therefore the total number of subjects analyzed for this outcome is less than the total number of subjects that comprise the SAS population.
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | Lisdexamfetamine Dimesylate (LDX) | Placebo
Number analyzed (Participants) | 59 | 58
Scores on a scale | -9.4 (14.43) | -5.9 (10.86)

14. Secondary Outcome: Change From Baseline in the Generalized Anxiety Disorder 7-Item (GAD-7) Total Score at Week 9, LOCF
Description: The GAD-7 is a 7-item self-report questionnaire for assessing anxiety severity. Each item is scored using a scale that ranges from 0 (not at all) to 3 (nearly every day) with total scores ranging from 0 to 21. Lower scores indicate a reduction in anxiety.
Time Frame: Baseline and week 9
Population: SAS
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | Lisdexamfetamine Dimesylate (LDX) | Placebo
Number analyzed (Participants) | 71 | 72
Scores on a scale | -4.4 (5.81) | -3.8 (5.43)

15. Secondary Outcome: Change From Baseline in Sheehan Suicidality Tracking Scale (STS) Total Score at Week 9
Description: The STS is an 8-question clinician-rated assessment of suicidal ideation, suicidal behavior, and accidents. The items are scored on a 5-point Likert scale from 0 (not at all) to 4 (extremely) and summed to produce a total score ranging from 0 to 32. Lower scores indicate reduced suicidal tendencies.
Time Frame: Baseline and week 9
Population: as for outcome 13
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | Lisdexamfetamine Dimesylate (LDX) | Placebo
Number analyzed (Participants) | 63 | 59
Scores on a scale | -0.1 (0.40) | 0.0 (0.13)

ADVERSE EVENTS:
Arm/Group | Lisdexamfetamine Dimesylate (LDX) | Placebo
Serious Adverse Events (participants affected / at risk) | 2/71 | 4/72
Other Adverse Events (participants affected / at risk) | 56/71 | 53/72
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Lisdexamfetamine Dimesylate (LDX) (N=71) | Placebo (N=72)
Loss of consciousness (Nervous system disorders) | 1 | 0
Suicidal ideation (Psychiatric disorders) | 1 | 0
Gastroenteritis (Infections and infestations) | 0 | 1
Rhabdomyolysis (Musculoskeletal and connective tissue disorders) | 0 | 1
Salmonellosis (Infections and infestations) | 0 | 1
Pelvic inflammatory disease (Infections and infestations) | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 2% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Lisdexamfetamine Dimesylate (LDX) (N=71) | Placebo (N=72)
Hyperacusis (Ear and labyrinth disorders) | 2 | 0
Abdominal pain (Gastrointestinal disorders) | 1 | 2
Constipation (Gastrointestinal disorders) | 2 | 0
Diarrhea (Gastrointestinal disorders) | 2 | 4
Dry mouth (Gastrointestinal disorders) | 11 | 6
Gastroesophageal reflux disease (Gastrointestinal disorders) | 0 | 3
Nausea (Gastrointestinal disorders) | 5 | 4
Vomiting (Gastrointestinal disorders) | 0 | 2
Fatigue (General disorders) | 4 | 4
Feeling jittery (General disorders) | 2 | 1
Irritability (General disorders) | 9 | 5
Nasopharyngitis (Infections and infestations) | 2 | 2
Sinusitis (Infections and infestations) | 1 | 4
Upper respiratory tract infection (Infections and infestations) | 6 | 4
Urinary tract infection (Infections and infestations) | 7 | 3
Viral infection (Infections and infestations) | 2 | 0
Blood pressure increased (Investigations) | 1 | 2
Heart rate increased (Investigations) | 3 | 0
Weight decreased (Investigations) | 2 | 0
Anorexia (Metabolism and nutrition disorders) | 2 | 1
Decreased appetite (Investigations) | 16 | 3
Back pain (Musculoskeletal and connective tissue disorders) | 3 | 1
Dizziness (Nervous system disorders) | 2 | 3
Headache (Nervous system disorders) | 16 | 11
Memory impairment (Nervous system disorders) | 2 | 0
Somnolence (Nervous system disorders) | 4 | 2
Tremor (Nervous system disorders) | 2 | 0
Abnormal dreams (Psychiatric disorders) | 2 | 1
Agitation (Psychiatric disorders) | 2 | 1
Anxiety (Psychiatric disorders) | 6 | 4
Insomnia (Psychiatric disorders) | 10 | 2
Nervousness (Psychiatric disorders) | 2 | 0
Sinus congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 2
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 4 | 0
Rash (Skin and subcutaneous tissue disorders) | 3 | 1
Uticaria (Skin and subcutaneous tissue disorders) | 2 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
If a multicenter publication is not submitted within twelve (12) months after conclusion, abandonment or termination of the Study at all sites, or after Sponsor confirms there shall be no multicenter Study publication, the Institution and/or such Principal Investigator may publish the results from the Institution site individually.